CLINICAL TRIAL: NCT00506051
Title: A Phase I, Open-Label Study to Assess the Safety and Tolerability of ZD6474 in Combination With Pemetrexed (Alimta) in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer After Failure of Prior Chemotherapy.
Brief Title: ZD6474(Vandetanib) + Alimta Combo Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00041
Record Dates: First submitted 2007-07-03; First posted 2007-07-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma; Non-Small Cell Lung; Lung Cancer
Keywords: Non-small cell lung cancer; lung cancer; alimta; vandetanib; phase 1
MeSH Terms: conditions — Carcinoma; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZD6474 (vandetanib) 100mg (Experimental)
  Interventions: Drug: ZD6474 (vandetanib) 100mg; Drug: pemetrexed
- ZD6474 (vandetanib) 300mg (Experimental)
  Interventions: Drug: pemetrexed; Drug: ZD6474 (vandetanib) 300mg

INTERVENTIONS:
Drug: ZD6474 (vandetanib) 100mg — once daily oral tablet
  Other Names: ZACTIMA™
  Arms: ZD6474 (vandetanib) 100mg
Drug: pemetrexed — intravenous infusion
  Other Names: Alimta®
Drug: ZD6474 (vandetanib) 300mg
  Other Names: ZACTIMA™
  Arms: ZD6474 (vandetanib) 300mg

SUMMARY:
The main purpose of this trial is to look to see if adding ZD6474 (100 mg or 300mg tablets) to Alimta chemotherapy in patients with non-small cell lung cancer is safe and will help control their symptoms and disease better than the chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced or metastatic non-small cell lung cancer
* Failure of first-line chemotherapy
* 1 or more measurable lesion by RECIST

Exclusion Criteria:

* Previous chemotherapy or radiotherapy within 4 weeks
* Significant cardiac events, arrythmias or other cardiac conditions
* Unacceptable laboratory measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To establish the safety & tolerability of ZD6474 when administered in combination w/Pemetrexed (Alimta) to patients w/locally advanced or metastatic NSCLC after failure of prior chemo, by assessment of AEs, vital signs, lab, ECG and physical exam. | assessed at each visit

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of ZD6474 and Pemetrexed when given in combination to patients with locally advanced or metastatic NSCLC after failure of prior chemotherapy, by assessment of appropriate pharmacokinetic (PK) parameters. | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

REFERENCES:
- [Background] de Boer R, Humblet Y, Wolf J, Nogova L, Ruffert K, Milenkova T, Smith R, Godwood A, Vansteenkiste J. An open-label study of vandetanib with pemetrexed in patients with previously treated non-small-cell lung cancer. Ann Oncol. 2009 Mar;20(3):486-91. doi: 10.1093/annonc/mdn674. Epub 2008 Dec 16. PMID 19088171
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1428&filename=CSR-D4200C00041.pdf
- See also: CSR-D4200C00041.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1428&filename=CSR-D4200C00041.pdf